CLINICAL TRIAL: NCT05047926
Title: Prehabilitation for Advanced Ovarian Cancer Patients
Brief Title: Prehabilitation for Stage IIIC-IV Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-005226; NCI-2021-09494 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Advanced Ovarian Carcinoma; Stage IIIC Fallopian Tube Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Primary Peritoneal Cancer AJCC v8; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Behavior Therapy; Exercise; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (surveys, CT, blood samples) (Experimental): Patients undergoing primary surgical intervention complete surveys, undergo CT, and undergo collection of blood samples at baseline.
  Interventions: Other: Survey Administration; Procedure: Computed Tomography; Procedure: Biospecimen Collection
- Cohort 2 (exercise, supplement, Resilient Living) (Experimental): Patients undergoing neoadjuvant chemotherapy complete physical activity for 30 minutes per day 3 times a week. Patients receive nutritional supplement drink up to 4.5 times daily, and complete Resilient Living program in-person or remotely over 60 minutes. Patients also undergo CT scans throughout the trial.
  Interventions: Dietary Supplement: Nutritional Supplement Drink; Other: Physical Activity; Other: Survey Administration; Procedure: Computed Tomography; Behavioral: Health Education
- Cohort 3 (exercise, supplement, coaching, Resilient Living) (Experimental): Patients undergoing neoadjuvant chemotherapy complete physical activity remotely for 30 minutes per day 3 times a week. Patients receive nutritional supplement drink up to 4.5 times daily. Patients also undergo health coaching remotely for 60 minutes weekly, complete Resilient Living program remotely over 60 minutes, and may wear a FitBit throughout the study.
  Interventions: Behavioral: Behavioral Counseling; Dietary Supplement: Nutritional Supplement Drink; Other: Physical Activity; Other: Survey Administration; Behavioral: Health Education; Other: Medical Device Usage and Evaluation

INTERVENTIONS:
Behavioral: Behavioral Counseling — Undergo behavioral counseling
  Other Names: Behavior Counseling; Behavioral Psychotherapy
  Arms: Cohort 3 (exercise, supplement, coaching, Resilient Living)
Dietary Supplement: Nutritional Supplement Drink — Given Boost or Ensure
  Other Names: Boost; Ensure; Polymeric Enteral Nutrition Formula
  Arms: Cohort 2 (exercise, supplement, Resilient Living); Cohort 3 (exercise, supplement, coaching, Resilient Living)
Other: Physical Activity — Complete physical activity assignments
  Arms: Cohort 2 (exercise, supplement, Resilient Living); Cohort 3 (exercise, supplement, coaching, Resilient Living)
Other: Survey Administration — Complete surveys
Procedure: Computed Tomography — Undergo CT scans
  Other Names: CAT; CAT Scan; Computed Axial Tomography (CAT); computerized axial tomography; Computerized axial tomography (procedure); Computerized Tomography (CT) scan; Computerized Tomography; CT; CT Scan; tomography
  Arms: Cohort 1 (surveys, CT, blood samples); Cohort 2 (exercise, supplement, Resilient Living)
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Cohort 1 (surveys, CT, blood samples)
Behavioral: Health Education — Complete Resilient Living program
  Arms: Cohort 2 (exercise, supplement, Resilient Living); Cohort 3 (exercise, supplement, coaching, Resilient Living)
Other: Medical Device Usage and Evaluation — Wear a FitBit
  Arms: Cohort 3 (exercise, supplement, coaching, Resilient Living)

SUMMARY:
This clinical trial evaluates whether a prehabilitation program started at the time of neoadjuvant chemotherapy will affect surgical recovery in patients with stage IIIC-IV ovarian, fallopian tube, or primary peritoneal cancer. A prehabilitation program may improve the quality of life after surgery for patients with ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the baseline difference in objective frailty measurements in patients with advanced ovarian cancer clinically deemed acceptable for primary surgery versus neoadjuvant chemotherapy.

II. To evaluate level of adherence and retention of patients with advanced ovarian cancer undergoing neoadjuvant chemotherapy with a prehabilitation program.

EXPLORATORY OBJECTIVE:

I. Will examine longitudinal trends and variability in function by the Short Physical Performance Battery (SPPB) over time and in response to the intervention.

OUTLINE: Patients are assigned to 1 of 3 cohorts.

COHORT 1: Patients undergoing primary surgical intervention complete surveys, undergo computed tomography (CT), and undergo collection of blood samples at baseline.

COHORT 2: Patients undergoing neoadjuvant chemotherapy complete physical activity for 30 minutes per day 3 times a week. Patients receive nutritional supplement drink up to 4.5 times daily, and complete Resilient Living program in-person or remotely over 60 minutes. Patients also undergo CT scans throughout the trial.

COHORT 3: Patients undergoing neoadjuvant chemotherapy complete physical activity remotely for 30 minutes per day 3 times a week. Patients receive nutritional supplement drink up to 4.5 times daily. Patients also undergo health coaching remotely for 60 minutes weekly, complete Resilient Living program remotely over 60 minutes, and may wear a FitBit throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Diagnosed with epithelial ovarian, fallopian tube, or primary peritoneal cancer based on imaging and physician diagnosis
* Suspected Stage IIIC or IV disease based on clinician staging and imaging
* Curative intent treatment with platinum-based chemotherapy
* Planned surgical intervention at some point during treatment course
* Ability to read English
* No diagnosed severe cognitive impairment
* Ability to provide consent
* Ability to utilize technology to watch online modules for the Resilient Living Program

Exclusion Criteria:

* Hemiplegia or paraplegia
* Current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Adherence to each prehabilitation component based on patient reported adherence (Cohorts 2 & 3) | Weekly up to 4 months
  Assessed based on patient reported adherence in Cohort 2. For cohort 3, adherence will be documented in MyDataHelps® and monitored remotely by the study team on the Care Evolution platform®. Participants will be evaluated weekly for compliance with the recommended exercise and nutrition and resilience interventions. Documentation of adherence will be through online patient messages, phone call, or during in person visits, whichever the patient prefers

SECONDARY OUTCOMES:
Implementation outcome | Up to 4 months
  Ability to recruit to this type of study and perform assessments at our institution will be measured based on the number of patients enrolled and the number of assessments completed throughout the study.
Difference in Short Physical Performance Battery (SPPB) at baseline between cohorts 1 and 2 | Baseline
  Short Physical Performance Battery (SPPB) will be measured at baseline in both cohorts.
Change of Short Physical Performance Battery (SPPB) over time in cohort 2 | Up to 4 months
  The Short Physical Performance Battery (SPPB) assessment will be administered and scored at baseline and at each study visit to assess lower extremity functioning (balance, gait, standing up from a chair).
Correlation of Short Physical Performance Battery (SPPB) to other assessments in cohorts 1 and 2 | Baseline, up to 4 months
  The following assessment tools will be completed at baseline, after chemotherapy/prior to surgery (cohort 2), 6 weeks post surgery (cohort 2), and after completion of all primary anti-cancer treatment (cohort 2): Short Physical Performance Battery (SPPB); gait speed (measured in meters/second); patient reported outcomes through Patient-Reported Outcomes Measurement Information System (PROMIS) short form surveys in the domains of pain, physical function, anxiety, emotional support, and fatigue; perceived stress scale; Fried Frailty index; body composition measurements on CT scans performed for clinical purposes; serum collection for frailty biomarker; and Mindfulness Attention awareness scale.
Correlation of assessments to compliance with interventions in cohort 2 | Baseline, up to 4 months
  The following assessment tools will be completed at baseline, after chemotherapy/prior to surgery (cohort 2), 6 weeks post surgery (cohort 2), and after completion of all primary anti-cancer treatment (cohort 2): Short Physical Performance Battery (SPPB); gait speed (measured in meters/second); patient reported outcomes through Patient-Reported Outcomes Measurement Information System (PROMIS) short form surveys in the domains of pain, physical function, anxiety, emotional support, and fatigue; perceived stress scale; Fried Frailty index; body composition measurements on CT scans performed for clinical purposes; serum collection for frailty biomarker; and Mindfulness Attention awareness scale.
Correlation of frailty assessments with clinical judgement of frailty | Baseline, up to 4 months
  The following assessments will be completed at baseline, after chemotherapy/prior to surgery (cohort 2), 6 weeks post surgery (cohort 2), and after completion of all primary anti-cancer treatment (cohort 2): Fried Frailty index; body composition measurements on CT scans performed for clinical purposes; serum collection for frailty biomarker; and Mindfulness Attention awareness scale. Results from these will be compared for correlation.
Correlation of body composition on computed tomography (CT) scans to frailty assessments | Baseline, up to 4 months
  The following assessments will be completed at baseline, after chemotherapy/prior to surgery (cohort 2), 6 weeks post surgery (cohort 2), and after completion of all primary anti-cancer treatment (cohort 2): Fried Frailty index; body composition measurements on CT scans performed for clinical purposes; serum collection for frailty biomarker; and Mindfulness Attention awareness scale. Results from these will be compared for correlation.
Qualitative outcomes of the facilitators, barriers, perceived benefits, and burdens | Baseline, up to 4 months
  Qualitative data from weekly contacts and exit interviews will be analyzed for codes and organized in themes to elucidate barriers, facilitators, perceived benefits, and negative effects of the program.
Acceptability of remote setting in Cohort 3 | 30 days
  Assessed using an Acceptability Questionnaire, which consists of 6 questions answered on a scale of 1-10 where 1=not at all and 10=extremely.

CONTACTS AND LOCATIONS:
Overall Officials: Amanika A. Kumar, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials